CLINICAL TRIAL: NCT00386945
Title: Tobacco Cessation Via Doctors of Chiropractic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA021349; 1R21DA021349-01 (NIH)
Record Dates: First submitted 2006-09-19; First posted 2006-10-12 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Tobacco Use Cessation
Keywords: Tobacco; Cessation.; Chiropractic patients.; Doctors of Chiropractic.; Health care providers.; Behavioral intervention.; Tobacco intervention.; Cigarettes.; Smokeless tobacco.; Smoking intervention.
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use | interventions — corticosteroid hormone-induced factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Non-Experiment Intervention consisting of an intervention based on the Clinical Practice Guideline: Treating Tobacco Use and Dependence and modified for use in chiropractic settings.
  Interventions: Behavioral: Brief counseling (Ask, Advise, Arrange)

INTERVENTIONS:
Behavioral: Brief counseling (Ask, Advise, Arrange) — Providers are trained to provide Ask, Advise and Arrange (brief cessation counseling) to all tobacco using patients. A Fax-to-Quit referral to a tobacco quit line and written materials on local cessation resources and pharmacotherapy are provided.

SUMMARY:
The purpose of the study is to develop an office-based tobacco intervention for chiropractic patients.

DETAILED DESCRIPTION:
Medical doctors, nurses, dentists, and dental hygienists have been shown to be effective in helping their patients quit tobacco. However, Doctors of Chiropractic (DCs) have not been utilized in this role. DCs can provide a unique channel for the conduct of tobacco interventions, but they currently receive little to no training in these techniques (Hawk & Evans, 2005). Doctors of Chiropractic are increasingly concerned with patients' use of cigarettes and smokeless tobacco. The chiropractic team provides educational and preventive services to patients, and the office visit can provide an extended opportunity to talk to patients about their tobacco use (Hawk, Long, Perillo, & Boulanger, 2004; Rupert, 2000). Given the health effects associated with chronic tobacco use, the chiropractic visit provides a "teachable moment" during which the DC can relate current health problems to tobacco use and provide brief counseling to patients who use tobacco (Gordon & Severson, 2001; Vogt, Lichtenstein, Ary, et al., 1989).

In the proposed developmental study, eight chiropractic clinics will participate in the design, implementation, and evaluation of an office-based tobacco cessation intervention. Adapted from previous office-based intervention protocols, the intervention will be based on Cognitive Learning Theory (Bandura, 1997) and the Clinical Practice Guidelines (Fiore, Bailey, Cohen, et al., 2000) and will also incorporate Motivational Interviewing techniques (Miller & Rollnick, 1991). Finally, using the RE-AIM framework (Glasgow, Vogt & Boles, 1999), we will assess individual-, clinic-, and organization-level variables that may affect the delivery of treatment for tobacco dependence, the implementation and maintenance of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Doctors of Chiropractic currently licensed by the Oregon Board of Chiropractic Examiners and actively engaging in patient care, their Chiropractic Assistants, and their Chiropractic patients who use tobacco

Exclusion Criteria:

* Chiropractic patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2006-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To design and refine our brief office-based tobacco intervention to use within chiropractic settings. | 12 months
To develop and refine study implementation protocols, DC and patient recruitment procedures, data collection strategies, and follow-up procedures. | 12 months
Prepare a working Manual of Procedures for a future randomized clinical trial. | 24 months

SECONDARY OUTCOMES:
Evaluate the reach of the intervention through an evaluation of the proportion of tobacco users of consenting age who give consent, the proportion who complete the baseline survey, and the reasons for not participating of those who decline. | 12 months
Evaluate the adoption of the intervention by interviewing clinic staff to identify the organizational-level factors that are related to participation. | 12 months
Assess the implementation of the intervention through an examination of patient report of receipt of the intervention components and change in providers' behavior and attitudes as a function of training. | 12 months
Explore the short-term maintenance of the intervention through an examination of change in provider behavior from baseline to 12 months after training and through an examination of change in clinic-level procedures. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Judith S. Gordon, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

REFERENCES:
- [Result] Gordon JS, Istvan J, Haas M. Tobacco cessation via doctors of chiropractic: results of a feasibility study. Nicotine Tob Res. 2010 Mar;12(3):305-8. doi: 10.1093/ntr/ntp203. Epub 2010 Jan 22. PMID 20097840